CLINICAL TRIAL: NCT00368082
Title: Administration of TGF-b Resistant LMP-Specific Cytotoxic T-Lymphocytes to Patients With Relapsed EBV-Positive Lymphoma
Brief Title: Autologous/Allogeneic TGFbeta-resistant LMP-specific CTL, Lymphoma (TGF-beta)
Acronym: TGF-beta
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: The Methodist Hospital Research Institute (Other); Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Helen Heslop, Professor, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17946-TGFBeta; TGF-beta (Other: Baylor College of Medicine); NCT00675571 (obsolete NCT alias)
Record Dates: First submitted 2006-08-22; First posted 2006-08-24 (Estimated); Last update posted 2025-10-31 (Actual); Status verified 2025-10

CONDITIONS: Lymphoma; Hodgkin's Disease; Relapse; Lymphoma, Non-Hodgkin
Keywords: EBV-Positive Lymphoma; Hodgkin´s Disease (HD); Non-Hodgkin's lymphoma (NHL); relapsed Hodgkin's disease; relapsed non-Hodgkin's disease; lymphoma; TGFbeta resistant LMP-specific CTLs; cytotoxic T cells
MeSH Terms: conditions — Lymphoma; Hodgkin Disease; Recurrence; Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- TGFbeta resistant LMP-specific CTLs (Experimental): CTLs be given by intravenous injection over 1-10 minutes through either a peripheral or a central line.
  If patients with active disease have stable disease or a partial response at their 6 week or subsequent evaluations they will be eligible to receive up to 6 additional doses of CTLs at 1-2 monthly intervals-each of which will consist of the same cell number as their second injection.
  Interventions: Biological: TGFbeta resistant LMP-specific CTLs

INTERVENTIONS:
Biological: TGFbeta resistant LMP-specific CTLs — Each patient will receive 2 injections, 14 days apart, according to the following dosing schedules:
  Group One:
  Day 0 2 x 10^7 cells/m2 Day 14 2 x 10^7 cells/m2
  Group Two:
  Day 0 6 x 10^7 cells/m2 Day 14 6 x 10^7 cells/m2
  Group Three:
  Day 0 1.5 x 10^8 cells/m2 Day 14 1.5 x 10^8 cells/m2
  Other Names: TGF-b Resistant LMP2A-Specific Cytotoxic T-Lymphocytes

SUMMARY:
Patients have a type of lymph gland cancer called HD, NHL or lymphoepithelioma (these 3 diseases will be referred to as "Lymphoma"). The lymphoma has come back or has not gone away after treatment. This is a research study using special immune system cells called TGFb-resistant LMP-specific cytotoxic T lymphocytes (DNR-CTL), a new experimental therapy.

Some patients with Lymphoma show signs of infection with the Epstein Barr virus (EBV) before or at the time of their Lymphoma diagnosis. EBV is found in the cancer cells of up to 1/2 the patients with Lymphoma, suggesting it may play a role in causing Lymphoma. The cancer cells infected by EBV are able to hide from the body's immune system and escape being killed by releasing a substance called Transforming Growth Factor-beta (TGFb). The investigators want to see if special white blood cells (called T cells) that have been given a gene that they hope will let them survive against TGFb and that have been trained to kill EBV infected cells can also survive in the blood and kill the tumor.

Investigators have used this sort of therapy with specially trained T cells to treat a different type of cancer that occurs after bone marrow and solid organ transplant called post transplant lymphoma. In this type of cancer they were able to successfully prevent and treat post transplant lymphoma. However when they used a similar approach in HD some patients had a partial response to this therapy, but no patients had a complete response. In a follow-up study they tried to find out if they could improve this treatment by growing T cells that recognize 2 of the proteins expressed on Lymphoma cells called LMP-1 and LMP2a. These special T cells were called LMP-specific cytotoxic T-lymphocytes (CTLs). Although some patients had tumor responses, CTL therapy alone did not cure those who had a lot of disease. Investigators think that a reason for this is that the tumor cells are releasing TGFb. For this reason, they want to find out if they can make the CTL resistant to TGFb by putting in a new gene called TGFb resistance gene. Investigators hope that this will improve this treatment for relapsed lymphoma. These TGFb-resistant LMP-specific CTLs are an investigational product not approved by FDA.

The purpose of this study is to find the largest safe dose of TGFb resistant LMP-specific CTLs, to learn what the side effects are and to see whether this therapy might help patients with Lymphoma.

DETAILED DESCRIPTION:
Investigators will test a biopsy of the tumor to see if the tumor cells are EBV positive and to see if the subject is eligible for this study. Then they will take some blood from the donor, which is used to grow T cells. First they will grow a special type of cell called dendritic cells (or monocytes), which stimulates the T cells and add a specially produced human adenovirus that carries the LMP1 and LMP-2a genes into the dendritic cells(or monocytes). Addition of a gene to the cells is known as gene transfer. These dendritic cells (or monocytes) are then used to stimulate T cells. The stimulation trains the T cells to kill cells with LMP on their surface. Investigators will then make more LMP-specific CTLs by stimulating them with EBV infected cells (which we will make from the subject's blood or the donor's blood by infecting them with EBV in the laboratory). They also will put the adenovirus that carries the LMP1 and LMP2 genes into these EBV infected cells so that they increase the amount of LMP1 and LMP2, which these cells have.

These EBV infected cells are treated with radiation so they cannot grow. Once sufficient numbers of T cells are made, investigators test them to see if they kill cells with LMP on their surface. To make sure that these cells won't attack the subjects tissues they test the cells against the skin cells or against T cells that they grow in the laboratory.

To make these CTL resistant to the effects of the TGFb released by the tumor we put in a new gene called a mutant TGFb receptor. Investigators used a mouse retrovirus that had been changed to stop it from causing infection to add the mutant TGFb receptor to the cells.

WHAT THE INFUSION WILL BE LIKE:

After the cells are made, they will be frozen. If the subject agrees to participate in this study, at the time they are scheduled to be treated, the cells will then be thawed and injected into the subject over 10 minutes.

Initially two doses of T cells will be given two weeks apart. If after the second infusion, there is a reduction in the size of the subject's lymphoma (or no increase) on CT or MRI scans as assessed by a radiologist, the subject can receive up to six additional doses if it would be to their benefit, if they would like to receive more doses, and if there is enough product remaining to give them additional doses.

This is a dose escalation study as investigators don't know what the highest dose of T cells with the new gene is safe. To find out, they will give the cells to 2 participants at one dose level. If that is safe they will raise the dose given to the next group of participants. The dose the subject will get will depend on how many participants get the agent before and how they react. The investigator will tell the subject this information.

All of the Treatments will be given by the Center for Cell and Gene Therapy at Texas Children's Hospital or Houston Methodist Hospital.

FOLLOW-UP STUDIES We will follow the subject after the injections. Total time participation for this study will be 15 years.

ELIGIBILITY:
INCLUSION CRITERIA:

1. Any patient, regardless of age or sex, with EBV-positive lymphoma, or lymphoepithelioma regardless of the histological subtype or EBV (associated)-T/NK-LPD all confirmed on any tissue sample.

   Primary refractory lymphoma or in second or subsequent relapse including after autologous or syngeneic stem cell transplant OR patients at a high risk for relapse defined as: (i) patients with primary refractory lymphoma or multiply relapsed lymphoma who are in remission but not eligible for autologous SCT or (ii) patients with relapsed lymphoma after autologous SCT who are in remission but not eligible for allogeneic SCT (Group A)

   OR

   Any patient who has received an allogeneic SCT for EBV Lymphoma or EBV (associated)-T/NK-LPD or Lymphoepithelioma (Group B)
2. Patients with life expectancy 6 weeks or greater from the time of CTL infusion.
3. Patients with a Karnofsky score of 50 or greater.
4. If post allogeneic SCT must not have less than 50% donor chimerism in either peripheral blood or bone marrow
5. Patients with bilirubin 3x normal or less, AST 5x normal or less, and Hgb greater than 8.0
6. Patients with a creatinine 2x normal for age or less
7. Patients with O2 saturations greater than 93% on room air (measured by pulse oximetry)
8. Patient, parent/guardian able to give informed consent.
9. Patients should have been off other investigational therapy for one month prior to entry in this study.

EXCLUSION CRITERIA:

1. Patients with a severe intercurrent infection.
2. Patients with evidence of GVHD greater than Grade II at time of enrollment.
3. HIV positive at time of procurement cells for CTL generation
4. Due to unknown effects of this therapy on a fetus, pregnant women are excluded from this research. The male partner should use a condom.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2006-04; Primary Completion 2013-09 (Actual); Study Completion 2031-07 (Estimated)

PRIMARY OUTCOMES:
Safety and MTD of 2 IV injections of autologous/syngeneic or allogeneic TGFb resistant LMP-specific cytotoxic T-lymphocytes. | 6 weeks
  Number of patients with Dose-Limiting Toxicity (DLT).

SECONDARY OUTCOMES:
Survival and immune function of TGFbeta-resistant LMP-specific cytotoxic T-lymphocytes. | 15 years
  Mean number of T cells transduced with vector.
Determine anti-viral and anti-tumor effects of TGFbeta resistant LMP-specific CTL. | 15 years
  Summarize tumor response by calculating overall response rates.

CONTACTS AND LOCATIONS:
Overall Officials: Helen E Heslop, MD, Principal Investigator — Baylor College of Medicine
Locations (2):
- United States (2):
  - Houston Methodist Hospital, Houston, Texas
  - Texas Childrens Hospital, Houston, Texas

REFERENCES:
- [Derived] Bollard CM, Tripic T, Cruz CR, Dotti G, Gottschalk S, Torrano V, Dakhova O, Carrum G, Ramos CA, Liu H, Wu MF, Marcogliese AN, Barese C, Zu Y, Lee DY, O'Connor O, Gee AP, Brenner MK, Heslop HE, Rooney CM. Tumor-Specific T-Cells Engineered to Overcome Tumor Immune Evasion Induce Clinical Responses in Patients With Relapsed Hodgkin Lymphoma. J Clin Oncol. 2018 Apr 10;36(11):1128-1139. doi: 10.1200/JCO.2017.74.3179. Epub 2018 Jan 9. PMID 29315015

DOCUMENTS (1):
  • Informed Consent Form (2018-08-21): https://cdn.clinicaltrials.gov/large-docs/82/NCT00368082/ICF_000.pdf